CLINICAL TRIAL: NCT07081282
Title: Precision Care Pathway Through Frailty and Cognitive Assessment Among Older Adults and Development of Care4Senior App, Intensive Aerobic Resistance Training and Brain Health Program in the Community
Brief Title: Precision Stratification for Frailty and Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Vivien Xi WU, PhD, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUS-IRB-2023-526
Record Dates: First submitted 2025-06-06; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Frailty; Cognitive Decline
MeSH Terms: conditions — Frailty; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Arm (Experimental): Participants will receive the CIRTAB intervention three times each week over 12-weeks.
  Interventions: Behavioral: Care4Senior mobile Application, Intensive Aerobic Resistance Training and Brain Health (CIRTAB)
- Active Control (Active Comparator): Participants will receive once in centre-based exercise health programme each week over 12-weeks.
  Interventions: Behavioral: Centre-Based Exercise Health Session
- Control (No Intervention): Participants will not participate in any exercise-related or brain health-related research studies or centre-based programme during trial period.

INTERVENTIONS:
Behavioral: Care4Senior mobile Application, Intensive Aerobic Resistance Training and Brain Health (CIRTAB) — Care4Senior mobile Application, Intensive Aerobic Resistance Training and Brain Health (CIRTAB)
  Other Names: CIRTAB
  Arms: Intervention Arm
Behavioral: Centre-Based Exercise Health Session — Participants will receive one time centre-based exercise health programme each week.
  Arms: Active Control

SUMMARY:
The Care4Senior mobile Application, Intensive Aerobic Resistance Training and Brain Health (CIRTAB) trial aim to test the effectiveness of an exercise, cognitive and lifestyle intervention amongst older adults over a 12-weeks trial period to prevent frailty and promote social bonding.

DETAILED DESCRIPTION:
In the Care4Senior mobile Application, Intensive Aerobic Resistance Training and Brain Health (CIRTAB) trial, participants will use the Care4Seniors 2.0 mobile application, in which physical and cognitive exercises will be provided to participants using this digital technology. Weekly in-person group exercise and cognitive sessions will also be conducted to prevent frailty, promote social bonding, as well as reduce social isolation and loneliness.

In the long term, this new service model has the potential to transform care, contain healthcare cost inflation and increase the efficiency of the lean manpower. It will translate knowledge into practice, resulting in impactful outcomes such as better self-management and healthy longevity. The CIRTAB program will raise the awareness of health behaviour, thus attracting more older adults to engage in preventive health and thus better prepare them for healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

1. Older Adults Aged 60 to 85 years old
2. Living in the community
3. Formally diagnosed with at least one chronic disease
4. Able to communicate in either English or Mandarin

Exclusion Criteria:

1. Severe vision or hearing impairment
2. Diagnosed with severe cognitive impairment (e.g. dementia)
3. Diagnosed with severe psychiatric disorders (e.g. psychotic disorders, major depressive disorder)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Frailty Status: - Edmonton Frailty Scale - Clinical Frailty Scale - Oral Frailty Index-8 | From enrollment to the end of treatment at 12 weeks.
  These measurements will be conducted by researchers at three timepoints - baseline, immediate post-intervention and 6 months post-intervention. The Edmonton Frailty Scale ranges from a minimum score of 0 (not frail) to a maximum score of 17 (severely frail), with higher scores indicating greater frailty.
  The Clinical Frailty Scale ranges from 1 (very fit) to 9 (terminally ill), with higher scores indicating greater frailty. The Oral Frailty Index-8 (OFI-8) ranges from a minimum score of 0 to a maximum of 8, with higher scores indicating greater oral frailty.
Presence of Sarcopenia: - Strength, Assistance with walking, Rise from a chair, Climb stairs, and Falls (SARC-F) Questionnaire | From enrollment to the end of treatment at 12 weeks.
  These measurements will be conducted by researchers at three timepoints - baseline, immediate post-intervention and 6 months post-intervention. The SARC-F Questionnaire ranges from a minimum score of 0 to a maximum of 10, with higher scores indicating greater risk of sarcopenia. A score of 4 or more suggests sarcopenia.
Presence of Cognitive Decline: - Montreal Cognitive Assessment - Symbol Digit Modalities Test - Cognitive Predictive Risk Score (developed from previous study) | From enrollment to the end of treatment at 12 weeks.
  These measurements will be conducted by researchers at three timepoints - baseline, immediate post-intervention and 6 months post-intervention. The Montreal Cognitive Assessment (MoCA) is a screening tool for mild cognitive impairment, scored out of 30 points, with higher scores indicating better cognitive function. The Symbol Digit Modalities Test (SDMT) assesses attention, processing speed, and visual-motor coordination, typically scored by the number of correct symbol-digit matches in 90 seconds, with higher scores indicating better performance. The total score for SDMT is 110. The Cognitive Predictive Risk Score developed from previous study stratify the participants into those with high risk of cognitive decline and those with low risk of cognitive decline.
Immunological Biomarkers: - C1q (complement component 1q) - IL-6 (Interleukin-6) | From enrollment to the end of treatment at 12 weeks.
  These measurements will be conducted by researchers at two timepoints - baseline and immediate post-intervention. The C1q levels typically range from 70 to 180 mg/L, with lower values indicating worsening immune function. The IL-6 levels normally range from 0 to 7 pg/mL, with higher values indicating increased inflammation.
Skeletomuscular Biomarkers: - IGF-1 (Insulin-like Growth Factor-1) - Myostatin | From enrollment to the end of treatment at 12 weeks.
  These measurements will be conducted by researchers at two timepoints - baseline and immediate post-intervention. The IGF-1 levels may range from 100 to 300 ng/mL, with lower levels associated with possible growth hormone deficiency. The Myostatin levels in serum range between 1 to 5 ng/mL, with higher levels associated with reduced muscle mass.

SECONDARY OUTCOMES:
Self-Care Ability - Self-Care of Chronic Illness Inventory (SCCII) | From enrollment to the end of treatment at 12 weeks.
  A generic measure designed to assess the process of self-care used by individuals with a variety of chronic conditions. It consists of 30 items that can be rated using 5-point Likert scale. There are four subdomains including self-help behavior, symptom management, health seeking behavior and self-care confidence. The minimum score is 28 and maximum score is 150. The higher the score, the better the self-care abilities.
Physical Activity Level - Global Physical Activity Questionnaire (GPAQ) | From enrollment to the end of treatment at 12 weeks.
  The GPAQ measures physical activity in Metabolic Equivalent of Task (MET) minutes per week, with 0 MET-minutes/week as the minimum (no activity) and no theoretical upper limit. The Global Physical Activity Questionnaire (GPAQ) does not have a fixed minimum or maximum score, the higher the GPAQ score, the greater the level of physical activity.
Physical Function - Short Physical Performance Battery (SPPB) | From enrollment to the end of treatment at 12 weeks.
  The SPPB is a standardised tool designed to assess lower limb function and overall physical performance in older adults. It has a minimum score of 0 and a maximum score of 12, with higher scores indicating better lower extremity function and physical performance.
Intrinsic Capacity - World Health Organization (WHO) Integrated Care for Older People (ICOPE) tool | From enrollment to the end of treatment at 12 weeks.
  The WHO ICOPE tool comprise nine domains test on cognitive decline, limited mobility, malnutrition, visual impairment, hearing loss, depressive symptoms, social care and support, carer support and urinary incontinence. Any failure or no to each domain will lead to a suggested pathway as per WHO. There is no fixed minimum or maximum scores, the lower the number of flagged areas, the better the intrinsic capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Active Ageing Centres Under Changi General Hospital's Community Health Team Cluster (East Region), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No